CLINICAL TRIAL: NCT02136368
Title: A Combined Exercise Program Plus Cognitive Training for Older Adults With Self-reported Cognitive Complaints: The Multi-modal, Mind-motor (M4) Study
Brief Title: Body and Brain Exercise for Older Adults With Memory Complaints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Rob Petrella, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: M4W18858
Record Dates: First submitted 2014-04-29; First posted 2014-05-13 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Cognitive Ability, General
Keywords: older adults; multiple-modality exercise; mind-motor exercise; self-reported cognitive complaints; global cognitive functioning; mobility; vascular function; sensorimotor function; brain imaging; community-based research; subjective cognitive complaints
MeSH Terms: interventions — Range of Motion, Articular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multi-Modal, Mind Motor Exercise (M4) (Experimental): Attend 60 minute exercise class three times per week for 24 weeks. Exercise class includes 45 minutes of multi-modal exercise and 15 minutes of mind-motor exercise.
  Interventions: Behavioral: Multi-modal exercise; Behavioral: Mind-Motor Exercise
- Multi-Modal Exercise (M2) (Active Comparator): Attend 60 minute exercise class three times per week for 24 weeks. Exercise class includes 45 minutes of multi-modal exercise and 15 minutes of balance and range of motion exercises.
  Interventions: Behavioral: Multi-modal exercise; Behavioral: Balance and range of motion exercises

INTERVENTIONS:
Behavioral: Multi-modal exercise — Community-based group exercise classes following Canadian Centre for Activity and Aging exercise guidelines. Exercise classes consist of 5 min warm-up, 20 min aerobic exercise, 5 min aerobic cool-down, 10 min full-body resistance exercise, 5 min stretching (total 45 min)
  Other Names: Exercise intervention
Behavioral: Mind-Motor Exercise — Square Step Exercise involves mimicking a stepping pattern demonstrated by an instructor. The stepping patterns become progressively difficult and involve forward, backward, lateral and diagonal movements on a 250cm long mat with 25cm square grids (15 min).
  Other Names: Square Stepping Exercise
  Arms: Multi-Modal, Mind Motor Exercise (M4)
Behavioral: Balance and range of motion exercises — Community-based group exercise designed to improve balance and range of motion of the joints (15 min)
  Arms: Multi-Modal Exercise (M2)

SUMMARY:
The purpose of this study is to investigate whether an exercise class with a cognitive (or brain) training component was more effective than a usual combined aerobic and resistance exercise class for older adults with cognitive complaints (such as concerns about changes in memory or thinking skills). It is hypothesized that the group randomized to the exercise class that includes additional brain training will have greater improvements in brain health.

DETAILED DESCRIPTION:
Older adults with self-reported cognitive complaints (CCs) may be at increased risk for the development of Alzheimer's disease and dementia. Cognitive decline in older adults, particularly reduced memory and executive function is associated with functional decline, institutionalization, and increased health care costs. Similarly, cardiovascular risk factors have been associated with cognitive and functional impairment in aging. Aerobic exercise has been shown to improve vascular function and blood flow in the brain's prefrontal cortex. In turn, resistance training can produce functional changes within distinct cortical regions during the encoding and recall of association tasks and has been shown to increase circulating neural growth factors (i.e., a proposed mechanism by which cognition may be preserved or improved in old age). Recent evidence also suggests that cognitive training may improve the cognitive performance of older adults.

Therefore, we will investigate the impact of a combined exercise program (multi-modality exercise; M2) compared to a combined exercise program with a cognitive component (multi-modality, mind-motor exercise; M4) on cognition, cognitive-motor, mobility, neural functioning and vascular outcomes in older adults with cognitive complaints. Community-based exercise programs for older adults provide widespread access, are relatively inexpensive, and provide opportunities for social interaction.

The primary purpose of this study is to compare the effects of the M2 and M4 exercise programs on brain health. This study will also examine the effects of the different exercise programs on cardiovascular risk factors and mobility. In a subset of participants, cognitive-motor and neural functioning outcomes will be examined.

ELIGIBILITY:
Inclusion Criteria:

* aged 55 years or older
* self-reported cognitive complaint (defined as answering yes to the question "Do you feel like your memory or thinking skills have gotten worse recently?).
* independent on instrumental activities of daily living

Exclusion Criteria:

* Probable Dementia (i.e., diagnosis OR Mini-Mental State Examination score <24)
* Other neurological conditions or major psychiatric disorders (i.e., Parkinson's disease; bipolar disorder)
* Previous history of severe cardiovascular conditions (i.e., myocardial infarction or stroke <1-year ago; end stage congestive heart failure; end stage renal disease)
* Severe sensory impairment (i.e., blind)
* Significant orthopedic conditions (i.e., severe osteoarthritis)
* Clinical depression (determined via >=16 on the Center for Epidemiologic Studies - Depression Scale AND review by primary study physician)
* Have blood pressure >180/100 mmHg or <100/60 mmHg
* Unable to comprehend questionnaire material
* Any other factors that could potentially limit ability to fully participate in the intervention

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Composite score from Cambridge Brain Sciences Cognitive Battery - 12 tasks | 6 months
  To assess global cognitive function

SECONDARY OUTCOMES:
Composite score from Cambridge Brain Sciences Cognitive Battery - 12 tasks | 12 months
  To assess global cognitive function
Gait variability (stride time) under dual-task conditions | 6 & 12 months
  Gait variability is the stride-to-stride fluctuations of the way someone walks and will be calculated as the coefficient of variation of step length (SD/mean x100). Measured with GAITRite system.
Gait variability (stride time) under single-task conditions | 6 & 12 months
  Gait variability is the stride-to-stride fluctuations of the way someone walks and will be calculated as the coefficient of variation of step length (SD/mean x100). Measured with GAITRite system.
Gait velocity (speed) under dual-task conditions | 6 & 12 months
  Average walking speed (gait velocity) measured with the GAITRite system
Gait velocity (speed) under single-task conditions | 6 & 12 months
  Average walking speed (gait velocity) measured with the GAITRite system
Step length (average) under dual-task conditions | 6 & 12 months
  Mean step length calculated from GAITRite system
Step length (average) under single-task conditions | 6 & 12 months
  Mean step length calculated from GAITRite system
Carotid Artery Compliance | 6 & 12 months
  Measured from non-invasive vascular assessment with B-mode Ultrasound over the carotid artery (in the neck).
Carotid Artery Intima-media thickness | 6 & 12 months
  Measured from non-invasive vascular assessment with B-mode Ultrasound over the carotid artery (in the neck).
Ambulatory Systolic Blood Pressure | 6 & 12 months
  Average systolic blood pressure over a 24 hour time period.
Clinic Systolic Blood Pressure | 6 & 12 months
  Average systolic blood pressure from in clinic final 2 (out of 3) readings
Ambulatory Diastolic Blood Pressure | 6 & 12 months
  Average diastolic blood pressure over a 24 hour time period.
Clinic Diastolic Blood Pressure | 6 & 12 months
  Average diastolic blood pressure from in clinic final 2 (out of 3) readings
Composite score of memory tasks from Cambridge Brain Sciences Cognitive Battery | 6 & 12 months
Composite score of executive function tasks from Cambridge Brain Sciences Cognitive Battery | 6 & 12 months
Composite score of concentration tasks from Cambridge Brain Sciences Cognitive Battery | 6 & 12 months
Total balance score | 6 & 12 months
  Total score calculated from the the Fullerton Advanced Balance scale

OTHER OUTCOMES:
Prosaccade reaction time in response to flash of light. | 6 months
  The reaction time of the eye when instructed to look toward a flash of light.
Change in blood flow to the pre-frontal cortex in response to a randomly selected cognitive task. | 6 months
  Neuroimaging assessment with functional magnetic resonance imaging
Antisaccade reaction time in response to flash of light. | 6 months
  The reaction time of the eye when instructed to look away from a flash of light.
Change in blood flow to the parietal cortex in response to a randomly selected cognitive task. | 6 months
  Neuroimaging assessment with functional magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Petrella, MD, PhD, Principal Investigator — The University of Western Ontario
Locations (1):
- Gymnasium, Woodstock, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boa Sorte Silva NC, Nagamatsu LS, Gill DP, Owen AM, Petrella RJ. Memory Function and Brain Functional Connectivity Adaptations Following Multiple-Modality Exercise and Mind-Motor Training in Older Adults at Risk of Dementia: An Exploratory Sub-Study. Front Aging Neurosci. 2020 Feb 25;12:22. doi: 10.3389/fnagi.2020.00022. eCollection 2020. PMID 32158386
- [Derived] Gregory MA, Gill DP, Shellington EM, Liu-Ambrose T, Shigematsu R, Zou G, Shoemaker K, Owen AM, Hachinski V, Stuckey M, Petrella RJ. Group-based exercise and cognitive-physical training in older adults with self-reported cognitive complaints: The Multiple-Modality, Mind-Motor (M4) study protocol. BMC Geriatr. 2016 Jan 16;16:17. doi: 10.1186/s12877-016-0190-9. PMID 26772171